CLINICAL TRIAL: NCT05974046
Title: A Phase I, Open Label Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of a Single Dose of Oral [14C]-IDV184001AN in Healthy Adult Male Participants
Brief Title: Single Dose Study of [14C]-IDV184001AN ([14C]-IDV184001) in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INDV-2000-105
Record Dates: First submitted 2023-06-06; First posted 2023-08-03 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder
Keywords: healthy volunteers; ADME; OUD; radiolabel; metabolism
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): [14C]IDV184001AN
  Interventions: Drug: [14C]IDV184001AN

INTERVENTIONS:
Drug: [14C]IDV184001AN — [14C]-IDV184001AN 200 mg/~100 µCi/ 15 g oral suspension
  Other Names: [14C]-IDV184001

SUMMARY:
The purpose of this open label study is to characterise the absorption, metabolism, excretion, and mass balance of [14C]-IDV184001AN ([14C]-IDV184001) in healthy adult male participants.

DETAILED DESCRIPTION:
The study is designed as an open label, single-dose study in healthy adult participants for the following reasons:

* Oral administration of IDV184001AN has demonstrated linear PK and thus [14C]IDV184001AN will be given as a single dose.
* A comparator is not necessary for the evaluation of the objectives.
* Blinding of the study treatment is not required as there is no comparator.
* Conducting the study in healthy participants mitigates the potential confounding effects of the disease state and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

  1. Participant must be 19 to 55 years of age inclusive, at the time of signing the informed consent.
  2. Participant must have body weight of a minimum of 50.0 kg at the Screening Visit and body mass index within the range 18.0 to 32.0 kg/m2 (inclusive).
  3. Participant must be male and who is healthy as determined by medical evaluation.
  4. Participant agrees to follow contraception guidelines from the time of dosing of study drug until at least 90 days after dosing of study drug. This includes use of highly effective contraception if sexually active with a non-pregnant partner of child-bearing potential, and agreement not to donate sperm from dosing until at least 90 days post-dose. There are no restrictions for a vasectomised male provided his vasectomy has been performed 4 months or more prior to dosing.
  5. Participant must be continuous non smoker who has not used nicotine and tobacco containing products for at least 3 months prior to dosing based on participant self-reporting.
  6. Participant must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and compliance with contraception guidelines.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. Have an ongoing medical history of clinically significant neurological, cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, psychiatric or other disorder as judged by an Investigator that could potentially affect the study outcomes or compromise participant safety.
  2. Have clinically significant abnormal biochemistry, haematology or urinalysis results as judged by an Investigator.
  3. Have a history of narcolepsy or sleep apnea.
  4. Have disorders that may interfere with drug absorption, distribution, metabolism and excretion processes.
  5. Current active hepatic or biliary disease.
  6. Participants with cholecystectomy <90 days prior to the Screening Visit.
  7. Positive test results for HIV-1/HIV-2 antibodies, HBsAg or Hepatitis C antibodies at the Screening Visit.
  8. Have a blood pressure reading outside of the following range: Systolic <86 or >149 mmHg; Diastolic <50 or >94 mmHg at the Screening Visit.
  9. Serious cardiac illness or other medical condition including, but not limited to:

     * Uncontrolled arrhythmias
     * History of congestive heart failure
     * QTcF >450 msec or history of prolonged QT syndrome
     * Myocardial infarction
     * Uncontrolled symptomatic angina
  10. History of suicidal ideation within 30 days prior to providing written informed consent as evidenced by answering "yes' to questions 4 or 5 on the suicidal ideation portion of the C-SSRS completed at the Screening Visit or history of a suicide attempt (per the C-SSRS) in the 6 months prior to informed consent.
  11. Healthy participants who are taking, or have taken, any prescribed or over the counter drugs (other than 2 grams of acetaminophen per 24-hour period as of Day 1 or thyroid hormone replacement therapy) or herbal remedies in the 14 days or 5 half-lives (whichever is longer) prior to dosing of study drug.
  12. Treatment with any known drugs that are moderate or strong inhibitors/inducers of CYP3A4 or CYP2C19, including St. John's Wort, within 30 days prior to dosing of study drug.
  13. Any consumption of food or drink containing poppy seeds, grapefruit or Seville oranges within 14 days prior to dosing of study drug.
  14. Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
  15. Positive test result for alcohol and/or drugs of abuse at the Screening Visit or at check-in.
  16. Concurrent treatment or treatment with an investigational drug or device within 30 days or 5 half-lives (whichever is longer) prior to dosing of study drug.
  17. Blood donation of approximately 500 mL or more within 56 days or plasma donation within 7 days prior to the Screening Visit.
  18. Known hypersensitivity to INDV-2000.
  19. Has less than 1 bowel movement every 2 days.
  20. Recent history of abnormal bowel movements, such as diarrhea, loose stools or constipation, within 2 weeks prior to dosing of study drug.
  21. Has received radiolabelled substances or has been exposed to radiation sources over the past 12 months or is likely to receive radiation exposure or radioisotopes within the next 12 months such that participation in this study would increase their total exposure beyond the recommended levels considered safe (ie, weighted annual limit recommended by the FDA 21CFR361 of 3000 mrem; FDA 2023).
  22. Site staff and/or participants who have a financial interest in, or an immediate family member of either the site staff and/or Indivior employees, directly involved in the study.
  23. Major surgical procedure (as defined by the Investigator) within 90 days prior to dosing of study drug or still recovering from prior surgery.
  24. Concurrent enrolment in another clinical study, unless it is an observational study.
  25. Participants who are unable, in the opinion of the Investigator, to comply fully with the study requirements.
  26. Any condition that, in the opinion of the Investigator or Indivior, would interfere with evaluation of the study drug or interpretation of participant safety or study results.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Director Clinical Development, Study Director — Indivior Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent of Radioactive Dose Excreted in the Urine, Feces, and Urine+Feces (%Dose) Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Percentage of total radioactivity recovered relative to dose (%Dose) in urine, feces and urine + feces (by time interval)
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Treatment
Number analyzed (Participants) | 7
Percentage of dose
  Urine, 0-4 hours post dose | 19.0 (25.9)
  Urine, 4-8 hours post dose | 25.3 (11.6)
  Urine, 8-12 hours post dose | 13.1 (18.2)
  Urine, 12-24 hours post dose | 13.5 (39.3)
  Urine, 24-48 hours post dose | 5.04 (48.6)
  Urine, 48-72 hours post dose | 0.941 (58.0)
  Urine, 72-96 hours post dose | 0.304 (55.0)
  Urine, 96-120 hours post dose | 0.150 (45.8)
  Urine, 120-144 hours post dose | 0.0919 (39.0)
  Urine, 144-168 hours post dose | 0.0585 (24.4)
  Feces, 0-24 hours post dose | 3.28 (6561.3)
  Feces, 24-48 hours post dose | 1.91 (707.0)
  Feces, 48-72 hours post dose | 0.892 (576.5)
  Feces, 72-96 hours post dose | 4.16 (380.2)
  Feces, 96-120 hours post dose | 1.16 (256.0)
  Feces, 120-144 hours post dose | 0.606 (303.4)
  Feces, 144-168 hours post dose | 0.292 (59.6)
  Urine+Feces, 0-4 hours post dose | 19.0 (25.9)
  Urine+Feces, 4-8 hours post dose | 25.3 (11.6)
  Urine+Feces, 8-12 hours post dose | 13.1 (18.2)
  Urine+Feces, 12-24 hours post dose | 18.3 (37.2)
  Urine+Feces, 24-48 hours post dose | 9.04 (70.6)
  Urine+Feces, 48-72 hours post dose | 1.87 (94.0)
  Urine+Feces, 72-96 hours post dose | 2.16 (534.2)
  Urine+Feces, 96-120 hours post dose | 1.34 (211.9)
  Urine+Feces, 120-144 hours post dose | 0.629 (313.7)
  Urine+Feces, 144-168 hours post dose | 0.318 (63.2)

2. Primary Outcome: Cumulative Percent of Radioactive Dose Excreted in the Urine, Feces, and Urine+Feces (Cum%Dose) Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Percentage of cumulative total radioactivity recovered relative to dose (Cum%Dose) in urine, feces, and urine+feces (0-168 hours)
Time Frame: Pre-dose to 168 hours post-dose
Measure: Mean (Standard Deviation); unit: Percent dose
Arm/Group | Treatment
Number analyzed (Participants) | 7
Percent dose
  Urine | 79.7 (5.769)
  Feces | 21.1 (5.342)
  Urine+Feces | 101 (0.6258)

3. Primary Outcome: Total Radioactivity AUClast in Plasma Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Total radioactivity pharmacokinetic parameter: AUC[last] (area under the concentration-time curve from time 0 to the time of the last quantifiable concentration calculated using the linear trapezoidal rule) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*h/mL
Arm/Group | Treatment
Number analyzed (Participants) | 7
ngEq*h/mL | 77300 (32.6)

4. Primary Outcome: Total Radioactivity AUClast in Whole Blood Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: as for outcome 3
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*h/g
Arm/Group | Treatment
Number analyzed (Participants) | 7
ngEq*h/g | 37700 (31.7)

5. Primary Outcome: Total Radioactivity AUC[0-∞] in Plasma Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Total radioactivity pharmacokinetic parameter: AUC[0-∞] (area under the concentration-time curve from time 0 extrapolated to infinite time) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*h/mL
Arm/Group | Treatment
Number analyzed (Participants) | 7
ngEq*h/mL | 83000 (33.4)

6. Primary Outcome: Total Radioactivity AUC[0-∞] in Whole Blood Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: as for outcome 5
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*h/g
Arm/Group | Treatment
Number analyzed (Participants) | 7
ngEq*h/g | 40100 (30.2)

7. Primary Outcome: Total Radioactivity AUC[Extrap(%)] in Plasma Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Total radioactivity pharmacokinetic parameter: AUC[extrap(%)] (percent of the area under the concentration-time curve due to extrapolation) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC extrapolated
Arm/Group | Treatment
Number analyzed (Participants) | 7
Percentage of AUC extrapolated | 6.84 (17.4)

8. Primary Outcome: Total Radioactivity AUC[Extrap(%)] in Whole Blood Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: as for outcome 7
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC extrapolated
Arm/Group | Treatment
Number analyzed (Participants) | 7
Percentage of AUC extrapolated | 5.60 (30.3)

9. Primary Outcome: Total Radioactivity Cmax in Plasma Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Total radioactivity pharmacokinetic parameter: Cmax (maximum observed concentration) as data permit. The Units of Measure for Cmax (i.e., " ngEq/mL") reflect the peak concentration that occurred from pre-dose to 168 hours post-dose.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL
Arm/Group | Treatment
Number analyzed (Participants) | 7
ngEq/mL | 6800 (16.5)

10. Primary Outcome: Total Radioactivity Cmax in Whole Blood Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Total radioactivity pharmacokinetic parameter: Cmax (maximum observed concentration) as data permit. The Units of Measure for Cmax (i.e., " ngEq/g)") reflect the peak concentration that occurred from pre-dose to 168 hours post-dose.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/g
Arm/Group | Treatment
Number analyzed (Participants) | 7
ngEq/g | 3980 (16.1)

11. Primary Outcome: Total Radioactivity Tmax in Plasma and Whole Blood Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Total radioactivity pharmacokinetic parameter: Tmax (time of Cmax) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Treatment
Number analyzed (Participants) | 7
hour
  Plasma | 2.01 (52.2)
  Whole blood | 1.94 (44.3)

12. Primary Outcome: Total Radioactivity λz in Plasma and Whole Blood Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Total radioactivity pharmacokinetic parameter: λz (terminal phase rate constant) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Treatment
Number analyzed (Participants) | 7
1/hour
  Plasma | 0.0180 (63.5)
  Whole blood | 0.0775 (46.3)

13. Primary Outcome: Total Radioactivity Ae[t1-t2] in Urine, Feces, and Urine+Feces Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Ae[t1-t2] (amount of total radioactivity excreted/recovered in urine, feces, and urine+feces within a given collection interval)
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mgEq
Arm/Group | Treatment
Number analyzed (Participants) | 7
mgEq
  Urine, 0-4 hour post dose | 38.8 (25.9)
  Urine, 4-8 hour post dose | 51.7 (11.7)
  Urine, 8-12 hour post dose | 26.8 (18.2)
  Urine, 12-24 hour post dose | 27.6 (39.3)
  Urine, 24-48 hour post dose | 10.3 (48.5)
  Urine, 48-72 hour post dose | 1.92 (58.0)
  Urine, 72-96 hour post dose | 0.620 (55.0)
  Urine, 96-120 hour post dose | 0.306 (45.6)
  Urine, 120-144 hour post dose | 0.188 (38.8)
  Urine, 144-168 hour post dose | 0.119 (24.3)
  Feces, 0-24 hour post dose | 6.69 (6587.9)
  Feces, 24-48 hour post dose | 3.89 (707.2)
  Feces, 48-72 hour post dose | 1.82 (575.4)
  Feces, 72-96 hour post dose | 8.50 (380.8)
  Feces, 96-120 hour post dose | 2.37 (255.7)
  Feces, 120-144 hour post dose | 1.24 (303.9)
  Feces, 144-168 hour post dose | 0.597 (59.5)
  Urine+feces, 0-4 hour post dose | 38.8 (25.9)
  Urine+feces, 4-8 hour post dose | 51.7 (11.7)
  Urine+feces, 8-12 hour post dose | 26.8 (18.2)
  Urine+feces, 12-24 hour post dose | 37.3 (37.3)
  Urine+feces, 24-48 hour post dose | 18.5 (70.4)
  Urine+feces, 48-72 hour post dose | 3.82 (93.9)
  Urine+feces, 72-96 hour post dose | 4.42 (535.1)
  Urine+feces, 96-120 hour post dose | 2.74 (211.6)
  Urine+feces, 120-144 hour post dose | 1.28 (314.2)
  Urine+feces, 144-168 hour post dose | 0.649 (63.1)

14. Primary Outcome: Total Radioactivity T1/2 in Plasma and Whole Blood Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: Total radioactivity pharmacokinetic parameter: T1/2 (apparent terminal half-life) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Treatment
Number analyzed (Participants) | 7
hour
  Plasma | 38.5 (63.5)
  Whole blood | 8.94 (46.3)

15. Primary Outcome: Total Radioactivity CumAe in Urine, Feces, and Urine+Feces Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: CumAe (cumulative amount of total radioactivity excreted/recovered in urine, feces, and urine+feces) (0-168 hour)
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mgEq
Arm/Group | Treatment
Number analyzed (Participants) | 7
mgEq
  Urine | 162 (7.4)
  Feces | 41.9 (26.1)
  Urine+feces | 206 (0.7)

16. Primary Outcome: Total Radioactivity CLr in Urine Following a Single Oral Dose of [14C]-IDV184001AN in Healthy Adult Male Participants
Description: CLr (renal clearance)
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Treatment
Number analyzed (Participants) | 7
L/hour | 2.10 (29.9)

17. Primary Outcome: Unlabeled IDV184001 and M12 AUC[Last] in Plasma Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: AUC[last] (area under the concentration-time curve from time 0 to the time of the last quantifiable concentration calculated using the linear trapezoidal rule) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment
Number analyzed (Participants) | 7
ng*h/mL
  Unlabeled IDV184001 plasma | 7150 (38.2)
  Unlabeled M12 plasma | 8940 (50.8)

18. Primary Outcome: Unlabeled IDV184001 and M12 AUC[0-∞] in Plasma Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: AUC[0-∞] (area under the concentration-time curve from time 0 extrapolated to infinite time) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment
Number analyzed (Participants) | 7
ng*h/mL
  Unlabeled IDV184001 in plasma | 7250 (37.3)
  Unlabeled M12 in plasma | 9070 (50.5)

19. Primary Outcome: Unlabeled IDV184001 and M12 AUC[Extrap(%)] in Plasma Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: AUC[extrap(%)] (percent of the area under the concentration-time curve due to extrapolation) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC extrapolated
Arm/Group | Treatment
Number analyzed (Participants) | 7
Percentage of AUC extrapolated
  Unlabeled IDV184001 in plasma | 0.775 (184.2)
  Unlabeled M12 in plasma | 1.08 (108.7)

20. Primary Outcome: Unlabeled IDV184001 and M12 Cmax in Plasma Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: Cmax (maximum observed concentration) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment
Number analyzed (Participants) | 7
ng/mL
  Unlabeled IDV184001 in plasma | 1380 (30.0)
  Unlabeled M12 in plasma | 1140 (32.0)

21. Primary Outcome: Unlabeled IDV184001 and M12 Tmax in Plasma Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: Tmax (time of Cmax) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Treatment
Number analyzed (Participants) | 7
hour
  Unlabeled IDV184001 in plasma | 1.43 (73.3)
  Unlabeled M12 in plasma | 2.29 (48.3)

22. Primary Outcome: Unlabeled IDV184001 and M12 λz in Plasma Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: λz (terminal phase rate constant) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Treatment
Number analyzed (Participants) | 7
1/hour
  Unlabeled IDV184001 in plasma | 0.277 (21.0)
  Unlabeled M12 in plasma | 0.172 (21.2)

23. Primary Outcome: Unlabeled IDV184001 and M12 T1/2 in Plasma Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: T1/2 (apparent terminal half-life) as data permit.
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Treatment
Number analyzed (Participants) | 7
hour
  Unlabeled IDV184001 in plasma | 2.50 (21.0)
  Unlabeled M12 in plasma | 4.02 (21.2)

24. Primary Outcome: Ratio of Unlabeled IDV184001 and M12 in Plasma to Plasma Total Radioactivity for AUC[Last] Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: Ratio of unlabeled IDV184001 and M12 in plasma to plasma total radioactivity for AUC[last] (area under the concentration-time curve from time 0 to the time of the last quantifiable concentration calculated using the linear trapezoidal rule), where appropriate
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio in plasma
Arm/Group | Treatment
Number analyzed (Participants) | 7
Ratio in plasma
  IDV184001 | 0.0926 (14.7)
  M12 | 0.120 (21.9)

25. Primary Outcome: Ratio of Unlabeled IDV184001 and M12 in Plasma to Plasma Total Radioactivity for Cmax Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: Ratio of unlabeled IDV184001 and M12 in plasma to plasma total radioactivity for Cmax (maximum observed concentration), where appropriate
Time Frame: Pre-dose to 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio in plasma
Arm/Group | Treatment
Number analyzed (Participants) | 7
Ratio in plasma
  IDV184001 | 0.202 (16.5)
  M12 | 0.173 (21.2)

26. Primary Outcome: Percentage of Total AUC of Each Identified Metabolite in Plasma Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: Determination of percentage of AUC (area under the concentration-time curve) of each identified metabolites to total AUC in plasma
Time Frame: Pre-dose to 168 hours post-dose
Measure: Number; unit: Percentage of AUC
Arm/Group | Treatment
Number analyzed (Participants) | 7
Percentage of AUC
  M12 | 23.6
  IDV184001 | 21.9
  M598 Isomer 1 | 15.5
  M422 Isomer 1 | 16.7
  M422 Isomer 2 | 13.7
  M275 Isomer 2 | 3.0
  M438 | 3.4
  M436 | 2.2

27. Primary Outcome: Percentage of Dose of Each Identified Metabolite in Urine Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: Determination of percentage of dose of each identified metabolites in urine
Time Frame: Pre-dose to 168 hours post-dose
Measure: Mean (Full Range); unit: Percentage of dose
Arm/Group | Treatment
Number analyzed (Participants) | 7
Percentage of dose
  M598 Isomer 1 | 21.9 [13.1 to 28.6]
  M436 | 8.2 [6.1 to 11.4]
  M275 Isomer 2 | 6.7 [5.4 to 8.3]
  M291, M275, and M289 Isomer 1 | 7.6 [4.9 to 10.8]
  M422 Isomer 1 and M628 Isomer 2 | 9.5 [7.0 to 12.3]

28. Primary Outcome: Percentage of Total AUC of Each Identified Metabolite in Feces Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: Determination of percentage of AUC (area under the concentration-time curve) of M436 metabolite to total AUC in feces
Time Frame: Pre-dose to 168 hours post-dose
Measure: Mean (Full Range); unit: Percentage of AUC
Arm/Group | Treatment
Number analyzed (Participants) | 7
Percentage of AUC | 14.7 [9.5 to 19.9]

29. Primary Outcome: Determination of the Ratio of Total Radioactivity Concentration Equivalents in Whole Blood Versus Plasma Following a Single Oral Dose of [14C] IDV184001AN in Healthy Adult Male Participants
Description: The ratio of total radioactivity concentration equivalents in whole blood relative to plasma at each time-matched determination of total radioactivity in whole blood and plasma
Time Frame: Pre-dose to 168 hours post-dose
Measure: Mean (Standard Deviation); unit: ml/g
Arm/Group | Treatment
Number analyzed (Participants) | 7
ml/g
  30 minutes post dose | 0.571 (0.06012)
  1 hour post dose | 0.567 (0.04071)
  2 hours post dose | 0.584 (0.02070)
  3 hours post dose | 0.574 (0.02637)
  4 hours post dose | 0.564 (0.01618)
  6 hours post dose | 0.574 (0.02699)
  8 hours post dose | 0.561 (0.05815)
  12 hours post dose | 0.573 (0.03147)
  24 hours post dose | 0.543 (0.03200)
  48 hours post dose | 0.219 (0.2734)
  72 hours post dose | 0.0750 (0.1837)
  96 hours post dose | 0 (0)
  120 hours post dose | NA (NA) — Not applicable as concentration was below the lower limit of quantification
  144 hours post dose | NA (NA) — Not applicable as concentration was below the lower limit of quantification
  168 hours post dose | NA (NA) — Not applicable as concentration was below the lower limit of quantification

30. Secondary Outcome: Assessment of the Safety and Tolerability (Incidence, Seriousness, Severity, and Relatedness of Treatment-emergent Adverse Events) of a Single Oral Dose of [14C] IDV184001AN as Determined by Adverse Event Reporting
Description: Incidence, seriousness, severity, and relatedness of treatment-emergent adverse events.
Time Frame: From informed consent signature to end of study (up to 11 days)
Population: Based on Guidance for Industry, Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials: 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Potentially life-threatening.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 7
Participants
  Any TEAE | 1
  Serious | 0
  Study-drug related | 1
  Serious and study drug-related | 0
  Severe | 0
  Toxicity Grade >= 3 | 0
  Resulted in study discontinuation | 0
  Resulted in death | 0

ADVERSE EVENTS:
Time Frame: From informed consent signature to end of study (up to 11 days).
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=7)
LACRIMATION INCREASED (Eye disorders) | 1
PHOTOPHOBIA (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT05974046/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT05974046/SAP_001.pdf